CLINICAL TRIAL: NCT04314921
Title: 10-week Yoga Practice Effect in Older Adults
Brief Title: 10-week Yoga Practice Effect on Cognitive and Motor Function in Older Adults
Acronym: BDNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LithuanianSportsU-3
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Aging; Healthy Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10-week Yoga (Experimental): Eighteen healthy elderly people, who were classified into two age groups, participated in this study. All participants had not practiced yoga before and were asked not to perform any sports activities while the research was ongoing. In the experimental group, participants (n = 18) had to participate in 10 weeks of yoga classes. In the control group, participants (n = 15) did not perform any exercises or other changes in their daily living life. All experimental group subjects participated in Himalayan yoga classes, which lasted 10 weeks: 2 times per week, 90 min per session. Yoga classes were conducted by 16-year-old qualified yoga instructor from Yoga Academy, Kaunas.
  Interventions: Other: Yoga trainings
- Control (No Intervention): In the control group, participants (n = 15) did not perform any exercises or other changes in their daily living life.

INTERVENTIONS:
Other: Yoga trainings — 10-week yoga sessions, 2 times per week, 90 min per session.
  Arms: 10-week Yoga

SUMMARY:
Thirty-three healthy elderly people, who were classified into two age groups, participated in this study. All participants had not practiced yoga before and were asked not to perform any sports activities while the research was ongoing. In the experimental group, participants (n = 18) had to participate in 10 weeks of yoga classes. In the control group, participants (n = 15) did not perform any exercises or other changes in their daily living life.

Experimental measurements: Brunel, PSS-14 and HAD questionnaires

ELIGIBILITY:
Inclusion Criteria:

* age, from 60 years old
* a statement by a local family physician about general good physical health
* never tired to practice yoga before

Exclusion Criteria:

* cardiovascular diseases
* musculoskeletal system diseases (osteoporosis, osteochondrosis, hernias)
* neurodegenerative diseases
* oncological diseases
* glaucoma
* injuries and surgeries in last 3 years

Ages: 60 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Brunel mood scale (BRUMS) | 10 weeks
  The Lithuanian translated version of the Brunel Mood Scale (BRUMS) was used in the present study. It was based on the originally developed to serve as a brief measure of mood before and after yoga intervention. The BRUMS (1) scale has 24 items arranged into six subscales: anger, confusion, depression, fatigue, tension and vigor. Each subscale has a numerical rating scale (0 = not at all, 1 = a bit, 2 = moderate, 3 = enough; 4 = extremely) from which research participant select the one best represents at that time. The results within subscale is summed and a score range from 0 to 16
Hospital anxiety and depression scale (HADS) | 10 weeks
  To determine the level of anxiety and depression of subjects was used HADS scale. The scale consists of totally 14 questions with the answers valued from 0 to 3. Half of questions addressed to estimate anxiety and rest - depression. The total scoring and conclusion for the both categories of questions: 0-7 = Normal; 8-10 = Borderline abnormal (borderline case); 11-21 = Abnormal (case)
Perceived stress scale -14 | 10 weeks
  The purpose of this scale is to assess the degree of stress in subjects' lives. It consists of questions about the frequency of feeling and thoughts during the past time period. Potential answers: 0-never; 1-almost never; 2-sometimes; 3-fairly often and 4-very often. The scores are obtained by reversing the scores on the four positive items: for example, 0=4, 1=3, 2=2, etc. and then summing across all items. Scores for the 14-item form range from 0 to 56, with higher scores indicating greater perceived stress
Human Free BDNF | 10 weeks
  Venous blood samples from median antecubital vein were collected in 5 ml vacuum tubes with a gel separator and was separated by centrifugation (15 min at 1200g) to make blood serum. Samples were aliquoted and stored at -800C until analysis. The serum concentration of Human Free BDNF was measured using an enzyme-linked immunoassay kit (R&D Systems, Minneapolis, USA)
Measurement of cognitive functions | 10 weeks
  Automated Neuropsychological Assessment Metrics Version 4 (ANAM-4; Vista Life, USA) was used to measure neurocognitive skills: mental flexibility, verbal working memory, inhibition control, visuospatial processing.
Psychomotor function evaluation | 10 weeks
  Participants were assessed by Dynamic Parameter Analyzer (DPA-1). Its measure motor functions: accuracy, reaction speed-accuracy.
Heart rate variability | 10 weeks
  R-R intervals were recorded using a Polar H7 sensor with a chest strap (Kempele, Finland).
Balance procedure | 10 weeks
  Postural sway activity was measured by a posturography method with a single piezoelectric force plate (Kistler, Slimline System 9286, Switzerland).

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian Sports Unviersity, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No